CLINICAL TRIAL: NCT04012151
Title: Arm and Finger Measurement for Blood Pressure Surveillance
Acronym: ARMFIN
Status: Active, not recruiting | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: ARMFIN; ANAESPRG19/012 (Other: SingHealth ANAES ACP)
Record Dates: First submitted 2019-05-27; First posted 2019-07-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Hypertension, Pregnancy-Induced
Keywords: Blood pressure measurement; Conicity index; Mid arm circumference; Cuff size
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant cohort: Parturients of gestational age >= 32 weeks will have measurements of arm length, MAC, proximal arm circumference, distal arm circumference, finger circumference to generate the conicity index.
  Interventions: Other: Physical measurement; Other: Cuff size fitting

INTERVENTIONS:
Other: Physical measurement — Parturients of gestational week >= 32 weeks will have their arms and fingers measured to generate the conicity index.
  Other Names: Measurement of fingers and arms
Other: Cuff size fitting — Fit on arm cuff and finger cuff as selected by investigators based on the measurement.
  Other Names: Cuff fitting for arm and finger

SUMMARY:
Accurate blood pressure (BP) measurement is critical in peripartum care. The cuff and bladder sizes affects the accuracy of BP measurement. Current international BP measurement recommendations are based on mid-arm circumference (MAC). However, evidence have shown the discrepancies between these sizes, leading to inaccuracy of BP measurement. This study will measure arm and finger size of 300 parturients in third trimester to determine whether the MAC, finger measurement or body mass index (BMI) is the best clinical predictor for non-standard cuff sizes for BP measurement.

DETAILED DESCRIPTION:
Accurate blood pressure (BP) measurement plays an important role in peripartum care as it is essential in detecting hypertensive disorders in pregnancy and medical decision making during the pregnancy. The cuff and bladder size have been highlighted as an important factor affecting the accuracy of BP measurement. Current international BP measurement recommendations are based on mid-arm circumference (MAC) assuming the arm is cylindrical in shape. However, evidence have shown a mismatch between these sizes, leading to BP overestimation or underestimation in obese patients. This is because the shape of the arm is a truncated cone instead of a cylinder, and the cuff will expand irregularly during inflation thus yielding inaccurate BP measurements. This is especially evident in Asian pregnant patients whereby no available guideline can recommend a suitable cuff for parturients with different MAC. Nexfin is a finger cuff device that can be a suitable alternative BP measurement device for such patients. In this study 300 parturients will be recruited in third trimester and undergoing nonemergent caesarean section in KKH. Patients' arm and finger sizes will be measured, and their user experience on current practices on BP measurement. The arm measurements will help to identify the proportion of women that may require non-standard cuff sizes for BP measurement. A conicity index will be determined whether the MAC, finger measurement or BMI is the best clinical predictor. The finger measurements will also help to determine the proportion of women that may require non-standard cuff sizes on the Nexfin device for BP measurement. The knowledge gathered in this pilot study will be used to design future studies in which the accuracy of Nexfin will be compared with standard BP measurement, which in turn will improve BP detection, subsequent patient monitoring and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists physical status 1 or 2 (ASA 1 or 2) parturients at 32 or more weeks of gestation
* Multiparous or nulliparous;
* Age 21-50 years old;
* Undergoing Caesarean section in our institution.

Exclusion Criteria:

* Emergent Caesarean section such that consent and measurements cannot be taken.

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant female in third trimester (>=32 weeks gestation)
Study Population: Pregnant women in Singapore
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Arm length (Left, Right) | During antenatal visit (1-2 hours). One visit only
  The distance (cm) between the tip of the acromion process to the tip of the olecranon process on the posterior aspect of the arm, with the elbow in the flexed position.
Mid Arm circumference (MAC)(Left, Right) | During antenatal visit (1-2 hours). One visit only
  The circumference (cm) of the arm at the mid-point of the arm length as measured above, with the arm hanging by the side.

SECONDARY OUTCOMES:
Proximal arm circumference (Left, Right) | During antenatal visit (1-2 hours). One visit only
  Arm circumference (cm) of the arm measured at the axilla, with the arm hanging by the side.
Distal arm circumference (Left, Right) | During antenatal visit (1-2 hours). One visit only
  The circumference (cm) at the elbow above the elbow crease, with the arm hanging by the side.
Finger circumference (Left, Right) | During antenatal visit (1-2 hours). One visit only
  The circumference (cm) of the mid-point of the middle phalanx of the middle finger will be measured with the hands placed flat on a table.
Feedback on experiences of previous BP measurement | During antenatal visit (1-2 hours). One visit only
  Participants will also respond to a three-point rating scale (Never, sometimes, always) about their experience of the procedures for previous BP measurement during the current pregnancy, with questions such as the length of time taken to obtain a reading, the need to change a cuff when taking BP, the need to take BP on the leg and whether the arm felt uncomfortable when taking blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Farida Ithnin, MMED (Anaes), Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Brien E, Asmar R, Beilin L, Imai Y, Mallion JM, Mancia G, Mengden T, Myers M, Padfield P, Palatini P, Parati G, Pickering T, Redon J, Staessen J, Stergiou G, Verdecchia P; European Society of Hypertension Working Group on Blood Pressure Monitoring. European Society of Hypertension recommendations for conventional, ambulatory and home blood pressure measurement. J Hypertens. 2003 May;21(5):821-48. doi: 10.1097/00004872-200305000-00001. No abstract available. PMID 12714851
- [Background] Pickering TG, Hall JE, Appel LJ, Falkner BE, Graves J, Hill MN, Jones DW, Kurtz T, Sheps SG, Roccella EJ. Recommendations for blood pressure measurement in humans and experimental animals: part 1: blood pressure measurement in humans: a statement for professionals from the Subcommittee of Professional and Public Education of the American Heart Association Council on High Blood Pressure Research. Circulation. 2005 Feb 8;111(5):697-716. doi: 10.1161/01.CIR.0000154900.76284.F6. PMID 15699287
- [Background] Perloff D, Grim C, Flack J, Frohlich ED, Hill M, McDonald M, Morgenstern BZ. Human blood pressure determination by sphygmomanometry. Circulation. 1993 Nov;88(5 Pt 1):2460-70. doi: 10.1161/01.cir.88.5.2460. No abstract available. PMID 8222141
- [Background] Brown MA, Lindheimer MD, de Swiet M, Van Assche A, Moutquin JM. The classification and diagnosis of the hypertensive disorders of pregnancy: statement from the International Society for the Study of Hypertension in Pregnancy (ISSHP). Hypertens Pregnancy. 2001;20(1):IX-XIV. doi: 10.1081/PRG-100104165. No abstract available. PMID 12044323
- [Background] Penaz J. Criteria for set point estimation in the volume clamp method of blood pressure measurement. Physiol Res. 1992;41(1):5-10. PMID 1610779
- [Result] Palatini P, Parati G. Blood pressure measurement in very obese patients: a challenging problem. J Hypertens. 2011 Mar;29(3):425-9. doi: 10.1097/HJH.0b013e3283435b65. No abstract available. PMID 21317721
- [Result] Fonseca-Reyes S, de Alba-Garcia JG, Parra-Carrillo JZ, Paczka-Zapata JA. Effect of standard cuff on blood pressure readings in patients with obese arms. How frequent are arms of a 'large circumference'? Blood Press Monit. 2003 Jun;8(3):101-6. doi: 10.1097/00126097-200306000-00002. PMID 12900586
- [Result] Bonso E, Saladini F, Zanier A, Benetti E, Dorigatti F, Palatini P. Accuracy of a single rigid conical cuff with standard-size bladder coupled to an automatic oscillometric device over a wide range of arm circumferences. Hypertens Res. 2010 Nov;33(11):1186-91. doi: 10.1038/hr.2010.146. Epub 2010 Aug 5. PMID 20686489
- [Result] Palatini P, Benetti E, Fania C, Malipiero G, Saladini F. Rectangular cuffs may overestimate blood pressure in individuals with large conical arms. J Hypertens. 2012 Mar;30(3):530-6. doi: 10.1097/HJH.0b013e32834f98a0. PMID 22278143
- [Result] Kho CL, Brown MA, Ong SL, Mangos GJ. Blood pressure measurement in pregnancy: the effect of arm circumference and sphygmomanometer cuff size. Obstet Med. 2009 Sep;2(3):116-20. doi: 10.1258/om.2009.090017. Epub 2009 Sep 1. PMID 27582825
- [Result] Eley VA, Roberts L, Rickards L, Pelecanos A, Blackie A, Zhang C, Christensen R, Barrett HL. Arm and finger measurements in the third trimester: Implications for blood pressure measurement. Pregnancy Hypertens. 2018 Oct;14:105-109. doi: 10.1016/j.preghy.2018.09.002. Epub 2018 Sep 5. PMID 30527095
- [Result] Wang J, Thornton JC, Russell M, Burastero S, Heymsfield S, Pierson RN Jr. Asians have lower body mass index (BMI) but higher percent body fat than do whites: comparisons of anthropometric measurements. Am J Clin Nutr. 1994 Jul;60(1):23-8. doi: 10.1093/ajcn/60.1.23. PMID 8017333
- [Derived] Lim MJ, Tan CW, Tan HS, Sultana R, Eley V, Sng BL. Correlation of patient characteristics with arm and finger measurements in Asian parturients: a preliminary study. BMC Anesthesiol. 2020 Aug 31;20(1):218. doi: 10.1186/s12871-020-01131-6. PMID 32867679

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT04012151/Prot_SAP_000.pdf